CLINICAL TRIAL: NCT05773274
Title: NET RETREAT: A Phase II Study of 177 Lutetium-DOTATATE Retreatment vs. Everolimus or Sunitinib or Cabozantinib in Metastatic/Unresectable Gastroenteropancreatic Neuroendocrine Tumours
Brief Title: Comparing Retreatment of 177Lu-DOTATATE PRRT Versus the Usual Treatment in Patients With Metastatic Unresectable Gastroenteropancreatic Neuroendocrine Tumors, NET RETREAT Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-00118; NCI-2023-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCTG-NE1 (Other: Canadian Cancer Trials Group); CCTG-NE1 (Other: CTEP); U10CA180863 (NIH)
Record Dates: First submitted 2023-03-16; First posted 2023-03-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Digestive System Neuroendocrine Tumor G1; Metastatic Digestive System Neuroendocrine Tumor G2; Unresectable Digestive System Neuroendocrine Tumor G1; Unresectable Digestive System Neuroendocrine Tumor G2
MeSH Terms: interventions — Specimen Handling; cabozantinib; Everolimus; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (177Lu-DOTATATE) (Experimental): Patients receive 177Lu-DOTATATE IV over 30 minutes Q8W. Treatment repeats for two cycles in the absence of disease progression or unacceptable toxicities. Patients also undergo CT scan and/or MRI and collection of blood samples while on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (everolimus) (Active Comparator): Patients receive everolimus PO QD, sunitinib PO QD or cabozantinib PO QD. Treatment continues in the absence of disease progression or unacceptable toxicities. Patients whose cancer worsens may cross over to ARM I. Patients also undergo CT scan and/or MRI and collection of blood samples while on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib; Procedure: Computed Tomography; Drug: Everolimus; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sunitinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib — Given PO
  Arms: Arm II (everolimus)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD-001; RAD001; Votubia; Zortress
  Arms: Arm II (everolimus)
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
  Arms: Arm I (177Lu-DOTATATE)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sunitinib — Given PO
  Arms: Arm II (everolimus)

SUMMARY:
This phase II trial compares the effect of retreatment with 177Lu-DOTATATE peptide receptor radionuclide therapy (PRRT) to the usual approach of treatment with everolimus, sunitinib, or cabozantinib in patients who have previously received 177Lu-DOTATATE for gastroenteropancreatic neuroendocrine tumor (GEPNET) that has spread from where it first started (primary site) to other places in the body (metastatic) and that cannot be removed by surgery (unresectable). PRRT is a type of radiation therapy for which a radioactive chemical is linked to a peptide (small protein) that targets tumor cells. When this radioactive peptide is injected into the body, it binds to a specific receptor found on some tumor cells. The radioactive peptide builds up in these cells and helps kill the tumor cells without harming normal cells. In this trial 177Lu-DOTATATE is used for PRRT. 177Lu-DOTATATE PRRT may increase the length of time until worsening of the GEPNET compared to the usual approach. Everolimus is in a class of medications called kinase inhibitors. It is also a type of angiogenesis inhibitor. Everolimus works by stopping tumor cells from reproducing and by decreasing blood supply to the tumor cells. Sunitinib and cabozantinib, block certain proteins, which may help keep tumor cells from growing. They may also prevent the growth of new blood vessels that tumors need to grow. Sunitinib malate is a type of tyrosine kinase inhibitor and a type of antiangiogenesis agent. Retreating with 177Lu-DOTATATE may work better than everolimus, sunitinib or cabozantinib in shrinking or stabilizing tumors in patients with metastatic and unresectable GEPNET who were previously treated with 177Lu-DOTATATE.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of lutetium Lu 177 dotatate (177Lu-DOTATATE) versus (vs.) everolimus or sunitinib (for pancreatic neuroendocrine [NET] patients only) or cabozantinib (United States [US] patients only) on progression-free survival (PFS) in patients with metastatic/unresectable GEPNET who have progressed following previous peptide receptor radionuclide therapy (PRRT).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity and safety of 177Lu-DOTATATE and everolimus or sunitinib (for pancreatic neuroendocrine NET patients only) or cabozantinib (US patients only).

II. To determine the effect of 177Lu-DOTATATE vs. everolimus or sunitinib (for pancreatic neuroendocrine NET patients only) or cabozantinib (US patients only) on overall response rate (ORR).

III. To evaluate the effect of 177Lu-DOTATATE vs. everolimus or sunitinib (for pancreatic neuroendocrine NET patients only) or cabozantinib (US patients only) on overall survival (OS).

IV. To evaluate post progression survival (PPS) and time to second objective disease progression (PFS2) for patients randomized to Arm 2 of the study and crossed over to Arm 1 at time of objective progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

V. To evaluate the effect of 177Lu-DOTATATE vs. everolimus or sunitinib (for pancreatic neuroendocrine NET patients only) or cabozantinib (US patients only) on patient quality of life (QoL).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive 177Lu-DOTATATE intravenously (IV) over 30 minutes every 8 weeks (Q8W). Treatment repeats for two cycles in the absence of disease progression or unacceptable toxicities. Patients also undergo computed tomography (CT) scan and/or magnetic resonance imaging (MRI) and collection of blood samples while on study.

ARM II: Patients receive everolimus orally (PO) on a daily basis (QD), sunitinib PO QD or cabozantinib PO QD. Treatment continues in the absence of disease progression or unacceptable toxicities. Patients whose cancer worsens may cross over to ARM I. Patients also undergo CT scan and/or MRI and collection of blood samples while on study.

After completion of study treatment, patients are followed up every 12 weeks until objective disease progression and then every 6 months until death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least >= 18 years of age
* Metastatic, histologically confirmed grade 1 or 2 well-differentiated gastroenteropancreatic neuroendocrine tumours, including NETs of unknown primary thought to be of gastroenterogancreatic origin, with positive Gallium-68 DOTATATE scan, Copper-64 DOTATATE scan or octreotide scan within the last 12 months is recommended but within the last 36 months is allowed. Lesions on Gallium-68 or Copper-64 DOTATATE scan or octreotide scan will be considered positive if the maximum standardized uptake value (SUVmax) of target lesion is > SUV mean of normal liver parenchyma

  * 7th Edition of the TNM Classification of Malignant Tumours
* Have received 3 or 4 cycles of PRRT using 177Lu-DOTATATE or a cumulative exposure of 22,200 MBq (600mCi) or 29,600 MBq (800 mCi) within +/- 10% variation within a 52-week period. No previous targeted alpha therapy is permitted
* Have had radiological progression per RECIST 1.1 after prior PRRT treatment and no sooner than 12 months from last scan performed post completion of initial PRRT where either stable disease, partial response, or complete response has been maintained throughout. Patients may have received previous systemic anti-cancer therapy subsequently, as long as they had benefited from initial PRRT for at least 12 months and have had confirmed progression per RECIST 1.1 on the intervening systemic anti-cancer therapy. Somatostatin analogues (SSA) administered for functional control are not considered an intervening systemic anti-cancer therapy. If intervening systemic anti-cancer therapy included a vascular endothelial growth factor (VEGF)-inhibitor, sunitinib can not be selected as standard of care on Arm 2. If intervening systemic anti-cancer therapy included an mammalian target of rapamycin (mTOR)-inhibitor, then everolimus can not be selected as the standard of care on Arm 2. If the intervening therapy is an alkylating agent, exposure of alkylating agent cannot exceed 12 months. The 12-month limit will also be applied to pre PRRT alkylator use as well
* Patients may have received previous ablative therapy or bland embolization as liver directed therapy however this must not have been received within 12 weeks from randomization date. Previous chemo and radio embolization are not permitted. Any lesion treated with an ablative technique as well as lesions in the lobe(s) of the liver treated with embolization shall not be included in target lesion assessment unless they have since progressed
* No ongoing toxicity from prior PRRT that is grade 3 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 80 g/L (>= 8.0 g/dL) (measured within 28 days prior to enrollment)
* Absolute neutrophil count >= 1.0 x 10^9/L (>= 1000/mm^3) (measured within 28 days prior to enrollment)
* Platelets >= 80 x 10^9/L (>= 80 x 10^3/mm^3) (measured within 28 days prior to enrollment)
* Total bilirubin < 1.5 x upper limit of normal (ULN) (upper limit of normal) (measured within 28 days prior to enrollment)

  * If confirmed Gilbert's, eligible providing =< 3.0 x ULN
* Creatinine clearance > 50 mL/min (measured within 28 days prior to enrollment)

  * Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft and Gault equation
* Prior or current use of somatostatin analogues is allowed for carcinoid syndrome control or in PRRT re-treatment patient population (Arm 1). Patients randomized to Arm 2 and receiving everolimus or sunitinib (pancreatic NET patients only) or cabozantinib (US patients only) will not be allowed to continue somatostatin analogues unless they have functional syndrome
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Males and females of reproductive potential must have agreed to use a highly effective contraceptive method during protocol treatment and for 7 months after the last dose of protocol treatment for females and 4 months after the last dose of protocol treatment for males. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. Men should avoid fathering a child for 4 months after the last dose of 177Lu-DOTATATE

  * Women of childbearing potential will have a pregnancy test to determine eligibility as part of the Pre-Study Evaluation; this may include an ultrasound to rule-out pregnancy if a false-positive is suspected. For example, when beta-human chorionic gonadotropin is high and partner is vasectomized, it may be associated with tumour production of human chorionic gonadotropin (hCG), as seen with some cancers. Patient will be considered eligible if an ultrasound is negative for pregnancy
* Patients must be accessible for treatment, response assessment, and follow up. Patients enrolled on this trial must be treated and followed at the participating center. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up

  * Patients must agree to return to their primary care facility for any adverse events which may occur through the course of the trial
* Patient must have access to everolimus or sunitinib (pancreatic NET patients only) or cabozantinib (US patients only). In the event that site/investigator is unable to provide access to the drug, patient will not be eligible for this trial
* Human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Major surgical procedures within 6 weeks from randomization date
* Known brain metastases, unless these metastases have been treated, stabilized and off steroids for at least 4 weeks prior to enrollment in the study. Patients with a history of brain metastases must have a head CT and/or MRI with contrast to document stable disease prior to enrollment in the study
* Uncontrolled congestive heart failure no worse than New York Heart Association Class (NYHA) IIB
* Inability to swallow oral medications or gastrointestinal disease limiting absorption of oral agents
* Patients with any other significant medical or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study
* Pregnant women are excluded from this study because 177Lu-DOTATATE is a peptide receptor radionuclide therapy with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 177Lu-DOTATATE, breastfeeding should be discontinued if the mother is treated with everolimus or sunitinib or cabozantinib (US patients only) and for 2.5 months following the last treatment with 177Lu-DOTATATE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to any documented evidence of tumour progression or death from any cause, assessed up to 3 years
  The PFS of patients of both treatment groups will be described by Kaplan-Meier method and the median PFS will be estimated using the same method. A one-sided stratified log-rank test adjusting for the stratification factor at randomization will be the primary method to compare the difference in PFS between the experimental and control treatments, at the 5% level. A stratified Cox model adjusting for duration of durable response to the initial peptide receptor radionuclide therapy (durable response >= 24 months versus [vs.] < 24 months) at randomization and with one single treatment covariate will be used to estimate the hazard ratio and associated one-sided 95% confidence interval. Sensitivity analysis adjusting for all three stratification factors at randomization will also be performed.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 3 years
  The OS of patients of both treatment groups will be described by Kaplan-Meier method and the median OS will be estimated using the same method. A one-sided stratified log-rank test adjusting for the stratification factor at randomization will be the primary method to compare the difference in OS between the experimental and control treatments, at the 5% level. A stratified Cox model adjusting for the stratification factor at randomization and with one single treatment covariate will be used to estimate the hazard ratio and associated one-sided 95% confidence interval.
Objective response rate (ORR) | Up to 3 years
  Defined as the proportion of patients with a documented complete response and partial response based on Response Evaluation Criteria in Solid Tumors 1.1. The primary estimate of ORR will be based on all patients randomized. A Cochran-Mantel-Haenszel test adjusting for the duration of durable response to the initial peptide receptor radionuclide therapy (durable response >= 24 months vs. < 24 months) at the time of randomization will be used to compare the objective response rates between two arms and sensitivity analysis adjusting for all three stratification factors at randomization will also be performed.
Post progression survival (PPS) | From objective progression on everolimus to objective progression or death from any cause after cross-over to receive 177Lu-DOTATATE, assessed up to 3 years
  Median PPS and associated two-sided 90% confidence interval will be estimated using the Kaplan-Meier method.
Time to second objective disease progression (PFS2) | From randomization to objective tumor progression or death from any cause after the cross-over, assessed up to 3 years
  Median PFS2 and associated two-sided 90% confidence interval will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Simron Singh, Principal Investigator — Canadian Cancer Trials Group
Locations (31):
- United States (26):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- Canada (5):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm